CLINICAL TRIAL: NCT02937168
Title: Distribution of Eosinophils in Asthma After Reslizumab (DEAR). A 7-Week, Placebo-Controlled, Double-Blinded, Parallel-Group, Imaging Study Using Positron Emission Tomography/Computer Tomography (PET/CT) to Characterize the Effect of Intravenous Reslizumab on Airway Inflammation in Patients With Eosinophilic Asthma
Brief Title: An Imaging Study Using PET/CT to Characterize the Effect of Intravenous Reslizumab on Airway Inflammation
Acronym: DEAR
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was terminated early due to challenges in recruitment. The decision to terminate the study was not related to any safety issues or concerns.
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C38072-AS-40105
Record Dates: First submitted 2016-10-14; First posted 2016-10-18 (Estimated); Results first posted 2019-08-06 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — reslizumab; Fluorodeoxyglucose F18

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Part 1: PET/CT Scan (Experimental): Healthy participants will have 2 PET/CT scan in Part 1: within 7 days of eligibility being confirmed, and 7 days after the first PET/CT scan. Participants will receive Fluorodeoxyglucose F-18 (FDG) as part of the PET/CT procedures and will provide sputum/blood samples.
  Interventions: Drug: Fludeoxyglucose F 18 (FDG)
- Part 2: Reslizumab (Experimental): Reslizumab 3.0 milligrams/kilogram (mg/kg) will be administered by intravenous (IV) infusion, over 20 to 50 minutes, at Baseline (Day 1) of Part 2. PET/CT scan will be done on Weeks 2, 4 and 6. Participants will receive FDG as part of the PET/CT procedures and will provide sputum/blood samples.
  Interventions: Drug: Reslizumab; Drug: Fludeoxyglucose F 18 (FDG)
- Part 2: Placebo (Placebo Comparator): Matching placebo will be administered by IV infusion at Baseline (Day 1) of Part 2. PET/CT scan will be done on Weeks 2, 4 and 6. Participants will receive FDG as part of the PET/CT procedures and will provide sputum/blood samples.
  Interventions: Drug: Fludeoxyglucose F 18 (FDG); Drug: Placebo

INTERVENTIONS:
Drug: Reslizumab — Reslizumab will be administered as per the dose and schedule specified in the arm.
  Arms: Part 2: Reslizumab
Drug: Fludeoxyglucose F 18 (FDG) — FDG will be administered by IV infusion prior to each PET/CT scan.
Drug: Placebo — Placebo matching to reslizumab will be administered as per the schedule specified in the arm.
  Arms: Part 2: Placebo

SUMMARY:
This is an exploratory study with the following primary objectives: 1) to establish that PET/CT of the lung can reliably distinguish healthy, non-asthmatic participants from participants with severe asthma and an eosinophilic phenotype and 2) to examine the utility of PET/CT for demonstrating that reslizumab produces a reduction in lung inflammation in participants with severe asthma and an eosinophilic phenotype .

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 through 50 years of age.
* Females that are either surgically sterile, are 2 years postmenopausal, or have a negative pregnancy test at screening.
* Females of childbearing potential (not surgically sterile or 2 years postmenopausal), have to use a medically accepted method of contraception and have to agree to continue to use of this method for the duration of the study and for 5 months after study drug administration.
* Participants with less that 10-pack year history of smoking.
* Have a previous diagnosis of asthma.
* Participants taking inhaled fluticasone at a dosage of at least 440 micrograms (mcg) daily, or equivalent.
* The participant's baseline asthma therapy must be stable for 30 days prior to screening and judged by their treating physician to be able to continue without dosage changes throughout the study.
* Participants with a blood eosinophil level of at least 400 cells/microliter (cells/μL) at screening. Participants with a blood eosinophil level below 400 cells/μL will be given 2 additional screening opportunities to determine blood eosinophil levels.

  * Additional criteria apply; please contact the investigator for more information.

Exclusion Criteria:

* Participants requiring treatment with oral, intramuscular, or IV corticosteroids within 6 weeks of the Part 1 baseline visit for an asthma exacerbation.
* Participants with any other confounding underlying lung disorder including but not limited to: bronchiectasis, chronic obstructive pulmonary disorder, smoking greater than or equal to (≥)10 pack year history, pulmonary fibrosis, emphysema, cystic fibrosis, and lung cancer.
* Participants diagnosed with diabetes mellitus.
* Participants with pulmonary conditions and blood eosinophilia other than eosinophilic asthma.
* Participants with clinically meaningful comorbidity that can interfere with the study schedule or procedures, or compromise the participant's safety.
* Participants that are current smokers (that is, have smoked within the last 12 months prior to screening).
* Participants using systemic immunosuppressive, immunomodulating, or other biologic agents (including, but not limited to, anti-IgE mAb, methotrexate, cyclosporin, interferon-α, or anti-tumor necrosis factor mAb) within 6 months prior to screening. Participants whose treatment with anti-IgE mAb therapy (omalizumab) is considered ineffective by their physician may be included as potential participants when:

  1. The omalizumab (Xolair) therapy has been discontinued.
  2. The participant's blood eosinophil level meets inclusion criteria.
* Participants who have previously received an anti-hIL-5 mAb (for example, reslizumab, mepolizumab [Nucala]) or anti-IL-5 receptor mAb (eg, benralizumab). Participants whose treatment with mepolizumab or benralizumab is considered ineffective by their physician may be included as potential participants when:

  1. The mepolizumab or benralizumab therapy has been discontinued.
  2. The participant's blood eosinophil level meets inclusion criteria.
* Participants who had concurrent infection or disease that may preclude assessment of active asthma.
* Participants with a history of concurrent immunodeficiency (human immunodeficiency virus or acquired immunodeficiency syndrome or congenital immunodeficiency).
* Participants that had an active parasitic infection within 6 months prior to screening.
* Participants with any disorder that may interfere with drug absorption, distribution, metabolism, or excretion (including gastrointestinal surgery).
* Known hypersensitivity to study drug or to FDG/contrast agents
* Treatment with metformin.
* Compromised renal function.

  * Additional criteria apply; please contact the investigator for more information.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2017-05-24 (Actual); Study Completion 2017-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (1):
- Teva Investigational Site 13808, New Brunswick, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study consisted of 2 parts: Part 1, a 21-day positron emission tomography (PET)/computed tomography (CT) screening period, and Part 2 (only participants with asthma), a 6-week double blind treatment/assessment period.
Pre-assignment Details: Participants with eosinophilic asthma were to be randomly assigned 1:1 in a double-blind fashion in Part 2 of the study to receive either placebo or reslizumab. Study was terminated prior to administration of reslizumab.
Groups:
- Part 1: PET/CT Scan: Healthy participants had 2 PET/CT scan in Part 1: within 7 days of eligibility being confirmed, and 7 days after the first PET/CT scan. Participants received Fluorodeoxyglucose F-18 (FDG) as part of the PET/CT procedures and provided sputum/blood samples.
- Part 2: Reslizumab: Reslizumab 3.0 milligrams/kilogram (mg/kg) was planned to be administered by intravenous (IV) infusion, over 20 to 50 minutes, at Baseline (Day 1) of Part 2. PET/CT scan was to be done on Weeks 2, 4 and 6.
- Part 2: Placebo: Matching placebo was planned to be administered by IV infusion at Baseline. (Day 1) of Part 2. PET/CT scan was to be done on Weeks 2, 4 and 6.
Period: PET/CT Screening Period (21 Days)
Arm/Group | Part 1: PET/CT Scan | Part 2: Reslizumab | Part 2: Placebo
Started | 5 | 0 | 0
Completed | 5 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Double-Blind Treatment Period (6 Weeks)
Arm/Group | Part 1: PET/CT Scan | Part 2: Reslizumab | Part 2: Placebo
Started (No participants were recruited for Part 2.) | 0 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All recruited healthy participants.
Groups:
- Part 1: PET/CT Scan: Healthy participants had 2 PET/CT scan in Part 1: within 7 days of eligibility being confirmed, and 7 days after the first PET/CT scan. Participants received FDG as part of the PET/CT procedures and provided sputum/blood samples.
Arm/Group | Part 1: PET/CT Scan
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.4 (10.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Average Global Lung Glycolysis (GLG) at Baseline (Day 1)
Description: GLG is the total FDG uptake in the whole lung. A region of interest (ROI) was drawn around lung boundary in each axial slice. Standardized uptake value (SUV) mean and area of each ROI was recorded. Using the formula: area*slice thickness the volume of each slice was calculated. Then the SUVmean of each slice was multiplied by the volume of the corresponding slice, which represented the total FDG uptake in one slice. This number for each slice was summed together to provide GLG of that lung. Average between GLG of right lung and GLG of left lung was reported.
Time Frame: Baseline (Day 1) of Part 1
Population: All recruited healthy participants.
Measure: Mean (Standard Deviation); unit: cubic centimeters (cm^3)
Arm/Group | Part 1: PET/CT Scan
Number analyzed (Participants) | 5
cubic centimeters (cm^3) | 668.08 (191.83)

2. Primary Outcome: Part 1: Average Global Lung Glycolysis (GLG) at Day 8
Description: GLG is the total FDG uptake in the whole lung. ROI was drawn around lung boundary in each axial slice. SUV mean and area of each ROI was recorded. Using the formula: area*slice thickness the volume of each slice was calculated. Then the SUVmean of each slice was multiplied by the volume of the corresponding slice, which represented the total FDG uptake in one slice. This number for each slice was summed together to provide GLG of that lung. Average between GLG of right lung and GLG of left lung was reported.
Time Frame: Day 8
Population: All recruited healthy participants.
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | Part 1: PET/CT Scan
Number analyzed (Participants) | 5
cm^3 | 621.71 (208.74)

3. Primary Outcome: Part 2: Change From Baseline to Week 4 in GLG
Time Frame: Baseline, Week 4
Population: Part 2 of the study was not conducted, hence this outcome measure was not analyzed.
Groups:
- Part 2: Reslizumab: Reslizumab 3.0 mg/kg was planned to be administered by IV infusion, over 20 to 50 minutes, at Baseline (Day 1) of Part 2. PET/CT scan was to be done on Weeks 2, 4 and 6.
Arm/Group | Part 2: Reslizumab | Part 2: Placebo
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Part 2: Change From Baseline to Week 4 in Lung Parenchyma (LP) SUV Mean
Time Frame: Baseline, Week 4
Population: Part 2 of the study was not conducted, hence this outcome measure was not analyzed.
Arm/Group | Part 2: Reslizumab | Part 2: Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Part 2: Change From Baseline to Week 4 in Blood Eosinophil Counts
Time Frame: Baseline, Week 4
Population: Part 2 of the study was not conducted, hence this outcome measure was not analyzed.
Arm/Group | Part 2: Reslizumab | Part 2: Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change From Baseline to Week 4 in Forced Expiratory Volume in 1 Second (FEV1)
Time Frame: Baseline, Week 4
Population: Part 2 of the study was not conducted, hence this outcome measure was not analyzed.
Arm/Group | Part 2: Reslizumab | Part 2: Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change From Baseline to Week 4 in Fractional Exhaled Nitric Oxide (FeNO)
Time Frame: Baseline, Week 4
Population: Part 2 of the study was not conducted, hence this outcome measure was not analyzed.
Arm/Group | Part 2: Reslizumab | Part 2: Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change From Baseline to Week 4 in Asthma Quality of Life Questionnaire (AQLQ) Score
Time Frame: Baseline, Week 4
Population: Part 2 of the study was not conducted, hence this outcome measure was not analyzed.
Arm/Group | Part 2: Reslizumab | Part 2: Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence that develops or worsens in severity during the conduct of a clinical study and does not necessarily have a causal relationship to the study drug. SAEs included death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized the participant and required medical intervention to prevent 1 of the outcomes listed in this definition. A summary of serious and non-serious AEs regardless of causality is located in 'Reported Adverse Events module'.
Time Frame: 21 days
Population: All recruited healthy participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: PET/CT Scan
Number analyzed (Participants) | 5
Participants
  Any AEs | 1
  SAEs | 0

ADVERSE EVENTS:
Time Frame: AEs were collected in Part 1 (21 days).
Description: All recruited healthy participants were analyzed.
Arm/Group | Part 1: PET/CT Scan
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 1/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: PET/CT Scan (N=5)
Right-hand injury (General disorders) | 1

LIMITATIONS AND CAVEATS:
The study was terminated early due to challenges in recruitment. The decision to terminate the study was not related to any safety issues or concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.

DOCUMENTS (2):
  • Study Protocol (2016-06-24): https://cdn.clinicaltrials.gov/large-docs/68/NCT02937168/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-30): https://cdn.clinicaltrials.gov/large-docs/68/NCT02937168/SAP_001.pdf